CLINICAL TRIAL: NCT00440908
Title: A Prospective Observational Cohort Study Tracking Laboratory Markers for Changes Over Time, After Converting Dialyzer Practice From Reuse to Single Use in Outpatient Dialysis Units
Brief Title: Inflammation and Nutritional Parameters in Hemodialysis Patients Using Reprocessed Dialyzers
Status: Completed | Type: Observational
Sponsor: Fresenius Medical Care North America (Industry)
Responsible Party: Raymond Hakim, MD PhD, Fresenius Medical Care North America
Other Study IDs: 07-032
Record Dates: First submitted 2007-02-26; First posted 2007-02-27 (Estimated); Last update posted 2008-05-07 (Estimated); Status verified 2008-05

CONDITIONS: End Stage Renal Disease; Inflammation
Keywords: Dialyzer reuse; Inflammatory markers; Nutritional status
MeSH Terms: conditions — Kidney Failure, Chronic; Inflammation

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The study is a prospective cohort trial utilizing sequential laboratory results from excess serum obtained from hemodialysis patients (acting as their own controls). The objective of this study is to determine the impact of converting from reuse to single use of dialyzers on specific markers of nutrition (pre-albumin) and inflammation (CRP) in hemodialysis patients followed over a period of 6-months after conversion. The Hypothesis is: Comparing values obtained at baseline to values at the end of 6-months after conversion from reuse to single use in the same patients:

1. In patients with baseline CRP > 5 mg/L: Mean decrease of 5 mg/L
2. In patients with baseline CRP < 5 mg/L: > 95% will remain < 5 mg/L
3. Mean serum pre-albumin levels will increase by at least 3 mg/dL. The study population will be drawn from ~2,900 patients that are currently undergoing hemodialysis in 48 dialysis units that have been identified as continuing to reuse dialyzers and specifically are using a peracetic acid-based disinfectant (Renalin®), as of February 1, 2007. These facilities will be scheduled to convert to single use of dialyzers between May and December, 2007. The selection of patients will depend solely on the facility conversion date, on a first-come, first-served basis. All patients within the dialysis facility that provide blood specimen for their routine monthly lab draws will be eligible. The facilities and patients will be enrolled consecutively until the desired sample size of approximately 2,500 patients is reached

DETAILED DESCRIPTION:
The proposed project is an ancillary quality improvement study that intends to prospectively track serum markers of inflammation (C-reactive protein or CRP) and nutrition (pre-albumin) at baseline (within 2-months before conversion from reuse to single use of dialyzers) and at the end of a 6-month follow-up period after the conversion, in maintenance hemodialysis patients. The first 2,500 patients from a potential pool of ~2,900 patients from 48 dialysis units that are scheduled to convert from reuse to single use of dialyzers, will be included in the study. Apart from routine monthly laboratory measurements, the investigators, in collaboration with Spectra Laboratories (central lab) will perform measurements of CRP and pre-albumin on the excess blood (after all the routine blood chemistries have been obtained) from the patients selected to be part of the study cohort. It is anticipated that the nature of this study as a quality improvement project, with no additional burden to the patients since tests will only be performed on excess blood from samples already sent to the laboratory, and the utilization of the information only in aggregate with no identifiable personal health information will allow for this study to proceed without the need for informed consent from each individual patient. It is hypothesized that the survival benefit that has been observed in some epidemiological studies (including the prior experience at Fresenius Medical Care, North America) may be accompanied by and/or the result of, reduced inflammation and/or improvement of nutritional status in patients that are converted from reuse to single use of dialyzers. The study will compare the difference between the values of CRP and pre-albumin separately, at baseline and at the end of 6-months after the conversion. CRP levels are expected to decline while pre-albumin are expected to increase during the follow-up period. Even with a 20% dropout rate, the study is expected to have >90% power to detect a change in CRP of >3 mg/L and >99% power to detect a similar change in pre-albumin. The patients in this study are only a subset of a larger epidemiological study that will examine the impact of converting from reuse to single use of dialyzers on patient survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing hemodialysis in 48 dialysis units that have been identified as continuing to reuse dialyzers processed with peracetic acid-based disinfectant (Renalin®), as of February 1, 2007.

Exclusion Criteria:

* Hemodialysis patients not currently reusing reprocessed dialyzers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients receiving dialysis in facilities where re-use of dialyzers processed with Renalin is practiced
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Actual)
Dates: Start 2007-03; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Hakim, MD, PhD, Principal Investigator — Fresenius Medical Care North America; Eduardo Lacson, MD, MPH, Study Director — Fresenius Medical Care North America
Locations (1):
- Fresenius Medical Care North America, Waltham, Massachusetts, United States

REFERENCES:
- [Background] Lowrie EG, Li Z, Ofsthun N, Lazarus JM. Reprocessing dialysers for multiple uses: recent analysis of death risks for patients. Nephrol Dial Transplant. 2004 Nov;19(11):2823-30. doi: 10.1093/ndt/gfh460. Epub 2004 Aug 17. PMID 15316099